CLINICAL TRIAL: NCT03678896
Title: Close Reading and Creative Writing - CrewD Program. An Alternative Educational Method for Group Care Intervention in Type 2 Diabetes Management. A Randomized Trial
Brief Title: Creative Writing for Type 2 Diabetes Management
Acronym: CrewD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao Protectora dos Diabeticos de Portugal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CrewD trial
Record Dates: First submitted 2018-09-10; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Diabetes
Keywords: Type II Diabetes; Educational methods; Disease self-management
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CrewD Program approach (Experimental): The aim was to increase education about the disease by using narrative skills through the CrewD Program. The sessions were conducted by two group leaders: a health professional and a literature professor manager of creative writing groups.
  Each session had a title, which parallels the classical structured educational approach (active comparator condition), which was known in advance by the subjects: a) Who I am in Diabetes?; b) Nutrition; c) The body where I live; d) Fears; e) Can attention change things?; and f) Roots.
  Team leaders directed a discussion of different texts used in the sessions with the participants focusing on their feelings and on how the texts relate to themselves and to their diabetes. Patients were encouraged to participate and freely express their opinion.
  Interventions: Behavioral: CrewD Program
- Classical structured education (Active Comparator): Each session was 90 minutes long, with a similar internal structure in all of them. Each session included the following topics: a) Chronic Disease; b) Nutrition; c) Exercise; d) Complications; e) Self-management; and f) Diabetic foot. The sessions were held in a large room, in which the seats were arranged in circle. Every session was chaired by two healthcare providers, who worked as group leaders.
  There was a different visual presentation in each session, with relevant theoretical information. A board with sheets of paper was available for use in the discussion along with brochures about the disease.
  Patients were encouraged to actively participate and take part in group-problem solving. Group leaders guided the discussion by asking questions and encouraging the discussion.
  Interventions: Behavioral: Classical structured education

INTERVENTIONS:
Behavioral: CrewD Program — The CrewD Program - Creative reading and writing in Diabetes Program - is a Diabetes self-management education and support program to help people with Diabetes coping with the disease.
  Arms: CrewD Program approach
Behavioral: Classical structured education — The Classical educational approach consists in an educational method based on the presentation of relevant theoretical information to help people with Diabetes coping with the disease.
  Arms: Classical structured education

SUMMARY:
This study is related to the development of a new model of Group Care for patients with Diabetes - the CrewD Program, incorporating close reading and creative writing in group education. A randomized trial was designed to evaluate this intervention.

DETAILED DESCRIPTION:
A structured educational model for type 2 diabetic patients using Group Care is currently being used in several institutions for help managing diabetes in these patients. In this study, this model was adjusted by introducing literary texts and using narrative skills. A randomized trial was designed to determine whether group dynamic strategies using narrative and reading produce the same positive outcomes as a conventional group approach. A total of 49 patients with type 2 Diabetes were randomized to two different Group Care dynamics, one "control group", with a classical structured educational approach and another, "intervention group", with close reading and creative writing. Evaluation included anthropometrical measures, A1c and questionnaires for psychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with type 2 diabetes of >1 year known duration, aged < 85 years were included in the intervention.

Exclusion Criteria:

* Patients that did not complete the four assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A1c levels at 6 months | Up to 6 months
  Hemoglobin A1c is measured in mmol/mol units.

SECONDARY OUTCOMES:
Change from baseline in weight at 6 months | Up to 6 months
  Weight is measured in Kg.
Change from baseline in fat mass at 6 months | Up to 6 months
  Fat mass is measured in Kg/m2
Change from baseline in waist circumference at 6 months | Up to 6 months
  Waist circumference is measured in cm
Change from baseline in self-reported quality of life at 6 months | Up to 6 months
  The Diabetes Quality of Life Questionnaire (DQOL) is a self-report scale to assess quality of life. This scale comprises 13 items that are grouped in 4 subscales: 1) satisfaction with treatment, 2) impact of treatment, 3) worry about the future effects of diabetes, and 4) worry about social/vocational issues. A total score may be also computed from the sum of the 13 items. Higher scores indicate poorer quality of life, ranging from 13 to 65.
Change from baseline in self-reported locus of control at 6 months | Up to 6 months
  Locus of control is measured using the Diabetes Specific Locus of Control Scale (DLOC), which is a self-report scale directed to diabetes patients. This scale comprises 13 items that are grouped in 3 subscales: 1) internal locus of control; 2) external locus of control; and 3) powerful other locus of control. Higher scores reflect higher locus of control in each of these dimensions.
Change from baseline in self-reported empathy at 6 months | Up to 6 months
  Empathy is measured using a questionnaire - Jefferson Scale of Physician Empathy (JSPE-R), which comprises 9 items. Self-reported empathy levels are measured through a total score that is derived from the sum of the 9 items. The total score range from 9 to 63, in which higher scores depict higher empathy levels.
Change from baseline in self-reported group satisfaction at 6 months | Up to 6 months
  Group satisfaction is measured using a questionnaire - Group Satisfaction Scale (GSS). The GSS assess 2 dimensions: 1) satisfaction with therapist subscale and 2) content/group process subscale. A total score may be also computed from the sum of the 12 items that comprise this scale. The scores range from 12 to 60, in which higher scores reflect higher satisfaction levels.
Change from baseline in self-reported health | Up to 6 months
  The 36-Item Short Form Survey is used to assess health perception. This scale comprises 36 items that are divided in 8 dimensions: 1) vitality; 2) physical functioning; 3) bodily pain; 4) general health perceptions; 5) physical role functioning; 6) emotional role functioning; 7) social role functioning; and 8) mental health. These subscales are transformed into a scale range from 0-100, in which lower scores indicate worse health perception.

CONTACTS AND LOCATIONS:
Overall Officials: João Raposo, M.D., Study Chair — Associacao Protectora dos Diabeticos de Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haas L, Maryniuk M, Beck J, Cox CE, Duker P, Edwards L, Fisher EB, Hanson L, Kent D, Kolb L, McLaughlin S, Orzeck E, Piette JD, Rhinehart AS, Rothman R, Sklaroff S, Tomky D, Youssef G; 2012 Standards Revision Task Force. National standards for diabetes self-management education and support. Diabetes Care. 2014 Jan;37 Suppl 1(Suppl 1):S144-53. doi: 10.2337/dc14-S144. No abstract available. PMID 24357210
- [Background] Chrvala CA, Sherr D, Lipman RD. Diabetes self-management education for adults with type 2 diabetes mellitus: A systematic review of the effect on glycemic control. Patient Educ Couns. 2016 Jun;99(6):926-43. doi: 10.1016/j.pec.2015.11.003. Epub 2015 Nov 22. PMID 26658704
- [Background] Trento M, Gamba S, Gentile L, Grassi G, Miselli V, Morone G, Passera P, Tonutti L, Tomalino M, Bondonio P, Cavallo F, Porta M; ROMEO Investigators. Rethink Organization to iMprove Education and Outcomes (ROMEO): a multicenter randomized trial of lifestyle intervention by group care to manage type 2 diabetes. Diabetes Care. 2010 Apr;33(4):745-7. doi: 10.2337/dc09-2024. Epub 2010 Jan 26. PMID 20103547
- [Background] Trento M, Tomelini M, Basile M, Borgo E, Passera P, Miselli V, Tomalino M, Cavallo F, Porta M. The locus of control in patients with Type 1 and Type 2 diabetes managed by individual and group care. Diabet Med. 2008 Jan;25(1):86-90. doi: 10.1111/j.1464-5491.2007.02319.x. PMID 18199135
- [Background] Charon R, Hermann N, Devlin MJ. Close Reading and Creative Writing in Clinical Education: Teaching Attention, Representation, and Affiliation. Acad Med. 2016 Mar;91(3):345-50. doi: 10.1097/ACM.0000000000000827. PMID 26200577
- [Background] Pennebaker JW. Putting stress into words: health, linguistic, and therapeutic implications. Behav Res Ther. 1993 Jul;31(6):539-48. doi: 10.1016/0005-7967(93)90105-4. PMID 8347112
- [Background] Frattaroli J. Experimental disclosure and its moderators: a meta-analysis. Psychol Bull. 2006 Nov;132(6):823-65. doi: 10.1037/0033-2909.132.6.823. PMID 17073523
- [Background] Ingersoll GM, Marrero DG. A modified quality-of-life measure for youths: psychometric properties. Diabetes Educ. 1991 Mar-Apr;17(2):114-8. doi: 10.1177/014572179101700219. PMID 1995281
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Hojat M, Gonnella J, Mangione S, Nasca T, Magee M. (2003). Physician empathy in medical education and practice: experience with The Jefferson Scale of Physician Empathy. Seminars in Integrative Medicine 2003; 1(1): 25-41.
- [Background] Ferraro LA, Price JH, Desmond SM, Roberts SM. Development of a diabetes locus of control scale. Psychol Rep. 1987 Dec;61(3):763-70. doi: 10.2466/pr0.1987.61.3.763. No abstract available. PMID 3438399
- [Background] Marshall LE, Serran G, Cameron C. The Group Satisfaction Scale. Rockwood Psychological Services & Royal Ottawa Health Care Group - STU 2010.
- [Background] Funnell MM, Brown TL, Childs BP, Haas LB, Hosey GM, Jensen B, Maryniuk M, Peyrot M, Piette JD, Reader D, Siminerio LM, Weinger K, Weiss MA. National Standards for diabetes self-management education. Diabetes Care. 2011 Jan;34 Suppl 1(Suppl 1):S89-96. doi: 10.2337/dc11-S089. No abstract available. PMID 21193633
- [Background] Funnell MM, Anderson RM. Patient empowerment: a look back, a look ahead. Diabetes Educ. 2003 May-Jun;29(3):454-8, 460, 462 passim. doi: 10.1177/014572170302900310. No abstract available. PMID 12854337
- [Background] Rosal MC, Ockene IS, Restrepo A, White MJ, Borg A, Olendzki B, Scavron J, Candib L, Welch G, Reed G. Randomized trial of a literacy-sensitive, culturally tailored diabetes self-management intervention for low-income latinos: latinos en control. Diabetes Care. 2011 Apr;34(4):838-44. doi: 10.2337/dc10-1981. Epub 2011 Mar 4. PMID 21378213
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Trento M, Passera P, Borgo E, Tomalino M, Bajardi M, Cavallo F, Porta M. A 5-year randomized controlled study of learning, problem solving ability, and quality of life modifications in people with type 2 diabetes managed by group care. Diabetes Care. 2004 Mar;27(3):670-5. doi: 10.2337/diacare.27.3.670. PMID 14988283